CLINICAL TRIAL: NCT02176668
Title: A Randomized, Open-label, Multiple-dose, Partial Crossover Study to Explore the Pharmacokinetics and the Pharmacodynamics of YH4808 New Formulation in Healthy Subjects
Brief Title: The Exploration for Pharmacodynamics and Pharmacokinetics of YH4808 New Formulation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: YH4808-111
Record Dates: First submitted 2014-06-11; First posted 2014-06-27 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2015-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Cohort1-YH4808 NF 100 (Experimental): 7 days repeat administration of YH4808 New Formulation 100mg after meal
  Interventions: Drug: YH4808 NF 100
- Cohort1-YH4808 OF 200 (Experimental): (Partial cross over design) 7 days repeat administration of YH4808 Old Formulation 200mg after meal, 4 Weeks of wash out period, 7 days repeat administration of YH4808 New Formulation 200mg after meal
  Interventions: Drug: YH4808 OF 200; Drug: YH4808 NF 200
- Cohort1-YH4808 NF 200 (Experimental): (Partial cross over design) 7 days repeat administration of YH4808 New Formulation 200mg after meal, 4 Weeks of wash out period, 7 days repeat administration of YH4808 Old Formulation 200mg after meal
  Interventions: Drug: YH4808 OF 200; Drug: YH4808 NF 200
- Cohort1-YH4808 NF 400 (Experimental): 7 days repeat administration of YH4808 New Formulation 400mg after meal
  Interventions: Drug: YH4808 NF 400
- Cohort2-YH4808 NF 100 (Experimental): 7 days repeat administration of YH4808 New Formulation 100mg before meal
  Interventions: Drug: YH4808 NF 100
- Cohort2-YH4808 NF 200 (Experimental): (Partial cross over design) 7 days repeat administration of YH4808 New Formulation 200mg before meal, 4 Weeks of wash out period, 7 days repeat administration of YH4808 Old Formulation 200mg before meal
  Interventions: Drug: YH4808 OF 200; Drug: YH4808 NF 200
- Cohort2-YH4808 OF 200 (Experimental): (Partial cross over design) 7 days repeat administration of YH4808 New Formulation 200mg before meal, 4 Weeks of wash out period, 7 days repeat administration of YH4808 Old Formulation 200mg before meal
  Interventions: Drug: YH4808 OF 200; Drug: YH4808 NF 200
- Cohort2-YH4808 NF 400 (Experimental): 7 days repeat administration of YH4808 New Formulation 400mg before meal
  Interventions: Drug: YH4808 NF 400
- Cohort3-YH4808 OF 200 (Experimental): (Partial cross over design)
  1. 7 days repeat administration of YH4808 Old Formulation 200mg before bed, 4 Weeks of wash out period, 7 days repeat administration of YH4808 Old Formulation 200mg before dinner
  2. 7 days repeat administration of YH4808 Old Formulation 200mg before dinner, 4 Weeks of wash out period, 7 days repeat administration of YH4808 Old Formulation 200mg before bed
  Interventions: Drug: YH4808 OF 200
- Cohort3-YH4808 OF 400 (Experimental): (Partial cross over design)
  1. 7 days repeat administration of YH4808 Old Formulation 400mg before bed, 4 Weeks of wash out period, 7 days repeat administration of YH4808 Old Formulation 400mg before dinner
  2. 7 days repeat administration of YH4808 Old Formulation 400mg before dinner, 4 Weeks of wash out period, 7 days repeat administration of YH4808 Old Formulation 400mg before bed
  Interventions: Drug: YH4808 OF 200

INTERVENTIONS:
Drug: YH4808 NF 100 — The number of times : multiple-dose Rout : oral administration
  Arms: Cohort1-YH4808 NF 100; Cohort2-YH4808 NF 100
Drug: YH4808 OF 200 — The number of times : multiple-dose Rout : oral administration
  Arms: Cohort1-YH4808 NF 200; Cohort1-YH4808 OF 200; Cohort2-YH4808 NF 200; Cohort2-YH4808 OF 200; Cohort3-YH4808 OF 200; Cohort3-YH4808 OF 400
Drug: YH4808 NF 200 — The number of times : multiple-dose Rout : oral administration
  Arms: Cohort1-YH4808 NF 200; Cohort1-YH4808 OF 200; Cohort2-YH4808 NF 200; Cohort2-YH4808 OF 200
Drug: YH4808 NF 400 — The number of times : multiple-dose Rout : oral administration
  Arms: Cohort1-YH4808 NF 400; Cohort2-YH4808 NF 400

SUMMARY:
The objective of this clinical trial is to explore pharmacodynamics and pharmacokinetics of YH4808 New Formulation in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. healthy adult age 20 to 55 over 55kg with ideal body weight(BMI) 18.5 ~ 25
2. Subject who has no congenital, chronic disease and disease symptoms in medical examination result
3. negative to Helicobacter pylori in 13C urea breath test
4. Subject who judged to be eligible according to various test results including laboratory test(serum test, hematologic/blood chemistry examination, urine test, etc.) and 12-lead ECG test performed within 4 weeks before the first IP administration.
5. Subject who agreed to maintain contraception and comply with medically verified contraception methods (including infertility)

Exclusion Criteria:

1. Subject who has history or presence of clinically significant disease in liver, kidney, nervous system, respiratory system, endocrine system, blood tumor, cardiovascular, reproductive, musculoskeletal system, mental disorder, ophthalmologic disease, and skin disease in investigator's judgement.
2. Subject who has history of surgical operation or disease related to gastrointestinal symptoms (e.g. crohn's diseas, ulcer, etc. except for appendectomy or simple hernia) which could have influence on the absorption of IP.
3. Subject who is hypersensitive to components contained in YH4808 and other drugs(aspirin, antibiotics, etc.)
4. pregnant or lactating woman.
5. Other exclusions apply.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The Cmax of YH4808 | Day 1(Day 35), Day 7(Day 41)
  Day 1(Day 35); predose, 11 times after dosing, Day 7(Day 41); predose, 13 times after dosing
The AUC0-24h of YH4808 | Day 1(Day 35), Day 7(Day 41)
  Day 1(Day 35); predose, 11 times after dosing, Day 7(Day 41); predose, 13 times after dosing
The AUC0-24h of M3 | Day 1(Day 35), Day 7(Day 41)
  Day 1(Day 35); predose, 11 times after dosing, Day 7(Day 41); predose, 13 times after dosing
The Cmax of M3 | Day 1(Day 35), Day 7(Day 41)
  Day 1(Day 35); predose, 11 times after dosing, Day 7(Day 41); predose, 13 times after dosing

SECONDARY OUTCOMES:
the arithmetic mean of 24h intragastric pH monitoring | Day 1(Day7)~Day2(Day8)
the median of 24h intragastric pH monitoring | Day 1(Day7)~Day2(Day8)
The Duration of stomach maintained over pH4 or 5 | Day 1(Day7)~Day2(Day8)

CONTACTS AND LOCATIONS:
Overall Officials: Min soo Park, Ph.D, M.D., Principal Investigator — Yonsei Medical Center Severance Hospital Clinical Trials Center
Locations (1):
- Yonsei Medical Center Severance Hospital Clinical Trials Center, Seoul, South Korea